CLINICAL TRIAL: NCT02966223
Title: A Study to Assess the Effect of Y-90 Therapy on Non-target/Background Liver
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor prematurely withdrew financial support.
Sponsor: Indiana University (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Mark Tann, Associate Professor of Radiology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RADY-BTG-TANN-HIDA/0603
Record Dates: First submitted 2016-11-08; First posted 2016-11-17 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: HCC; Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRI and HIDA scan (Experimental)
  Interventions: Radiation: MRI and HIDA scan

INTERVENTIONS:
Radiation: MRI and HIDA scan — Pre y90 therapy each subject will undergo a HIDA and MRI scan. 3 months post Y90 - Each subject will undergo a second HIDA scan and MRI scan

SUMMARY:
The primary question of interest is quantifying the relationship between Y-90 liver therapy and liver damage. Little is known on this subject. Present assumptions and calculations of Y-90 administration are based on surgical lobar hepatectomies and external radiation beam therapies. The investigators hope that by using a functional model of the liver, the investigators can improve this important knowledge gap.

The investigators will be enrolling patients planning to receive Y-90 therapy for the treatment of liver malignancies. The diagnosis of a primary liver cancer, hepatocellular carcinoma (HCC), is usually made by a combination of specific imaging findings and clinical criteria; only rarely is a confirmatory biopsy performed. This is due to the high accuracy of the present diagnostic model and the significant risk of biopsy and tumor seeding.

Y-90 therapy involves administering radioactive particles to liver tumors by placing a catheter in a hepatic artery supplying the tumor using angiographic techniques and injection of these particles.

Y-90 Positron Emission Tomography-Computed Tomography (PET/CT) imaging has been established as a method to validate and quantitate distribution of Yttrium after Y-90 administration. The post Y-90 therapy PET/CT images provide an imaging distribution of the Y-90, which is essential for validation of administered versus planned dose to the liver lesion and background liver.

If the investigators can compare the Y-90 distribution to estimate background liver radiation distribution and dose (generated by the Y-90 PET/CT scan) combined with the global and regional function map (generated by the hepatobiliary [HIDA] scan performed before and after therapy), then the investigators will be assuming that the difference pre and post therapy in global and regional function can be ascribed to the Y-90 administration. The investigators will also analyze the Magnetic Resonance Imaging (MRI) and CT sets performed before and after therapy and correlate the imaging results collected with clinical findings such as ascites/encephalopathy and routine serological markers (bilirubin, albumin, International normalized ratio [INR], etc.). With this information, the investigators will have the potential to establish whether there is a relationship between Y-90 distribution to non-tumoral (normal) hepatic parenchyma and the incidence and severity of Radioembolization-Induced Liver Disease (REILD). This would have the potential to improve selection criteria and outcomes in populations selected for Y-90 therapy in the future.

DETAILED DESCRIPTION:
Little is known on the potential relationship between Y-90 liver therapy and liver damage this subject. Present assumptions and calculations of Y-90 administration are based on surgical lobar hepatectomies and external radiation beam therapies.

As most participants that need Y90 based liver therapies have compromised livers, the importance of knowing what potential collateral liver damage could be induced by Y90 is key so as not induce liver failure. Successful treatment of a liver malignancy would not be important if the potential mortality/morbidity risk of the treatment is higher or equal to the existing malignancy.

As apposed to anatomical imaging looking for changes in size/shape which are late changes, the investigators hope that by using a functional model of the liver, which can show early changes of liver damage, the investigators can improve the sensitivity for detection of liver damage and bridge this important knowledge gap. Additionally due to compensatory hypertrophy of the non treated liver, potential liver damage estimated by lab tests may be masked, again this emphasizes the importance of the measurement of the functional approach before and after therapy.

The investigators will be enrolling participants planning to receive Y-90 therapy for the treatment of liver malignancies. The diagnosis of a primary liver cancer, hepatocellular carcinoma (HCC), is usually made by a combination of specific imaging findings and clinical criteria; only rarely is a confirmatory biopsy performed. This is due to the high accuracy of the present diagnostic model and the significant risk of biopsy and tumor seeding.

Y-90 therapy involves administering radioactive particles to liver tumors by placing a catheter in a hepatic artery supplying the tumor using angiographic techniques and injection of these particles.

Y-90 PET/CT imaging has been established as a method to validate and quantitate distribution of Yttrium after Y-90 administration. The post Y-90 therapy PET/CT images provide an imaging distribution of the Y-90, which is essential for validation of administered versus planned dose to the liver lesion and background liver.

The investigators will be performing both specialized nuclear medicine HIDA and MRI scans aimed at constructing a functional map of the liver before and 3 months after therapy.

The investigators will compare the Y-90 distribution to estimate background liver radiation distribution and dose (generated by the Y-90 PET/CT scan) combined with the global and regional function map (generated by the HIDA and MRI scans performed before and after therapy), then the investigators will be assuming that the difference pre and post therapy in global and regional function can be ascribed to the Y-90 administration.

The investigators will also analyze the MRI and NM data sets performed before and after therapy and correlate the imaging results collected with clinical findings such as ascites/encephalopathy and routine serological markers (bilirubin, albumin, INR, etc.).

With this information, the investigators will have the potential to establish whether there is a relationship between Y-90 distribution to non-tumoral (normal) hepatic parenchyma and the incidence and severity of REILD. This would have the potential to improve selection criteria and outcomes in populations selected for Y-90 therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have the ability to understand and the willingness to sign a written informed consent document.
2. Subjects must be ≥ 18 years of age at the time of signing informed consent.
3. Subjects must have a diagnosis of hepatocellular carcinoma (HCC) and a treatment plan to undergo radioembolization therapy with Y-90 at Indiana University Health Hospital.
4. Subjects must be willing and able to comply with all procedures and visits required for this protocol (pre-treatment, during treatment, and post-treatment).

Exclusion Criteria:

1. Subjects who have contraindications for receiving Y-90 therapy and any routine procedures and imaging associated with Y-90 therapy, including subjects who are pregnant or are planning to become pregnant, will not be eligible to participate in this study. Female subjects who are of childbearing potential should inform her treating physician should she become pregnant at any time during the course of the study.
2. Subjects with contraindications for receiving hepatobiliary scans (HIDA scans) and Magnetic Resonance Imaging (MRI scans) will not be eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Tann, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI and HIDA Scan
Started | 20
Completed | 5
Not Completed | 15
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The trial was halted prematurely because sponsor withdrew funding. There is insufficient data to analyze. Inclusion criteria to participate in study being 18 years of age and older, Hepatocellular Carcinoma diagnoses and treatment plan to undergo radioembolization Y90 therapy, and not pregnant or planning to become pregnant during study.
Arm/Group | MRI and HIDA Scan
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants] — Average age of enrolled subjects is 66 years old.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] — Measure Description: Average age of enrolled population 66 years old. Average age of subjects who completed study 65 years old.
  years | 66 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of subjects that enrolled in study.
  Participants
    Female | 3
    Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Enrollment took place in Indianapolis, IN.
  Participants
    United States | 20
Enrollment [Count of Participants; unit: Participants] — Recruitment of volunteers who consented to participate in study.
  Participants | 20

OUTCOME MEASURES:

1. Primary Outcome: Primary
Description: Difference in regional liver function between pre and 3 months post Yttrium 90 delivery using the HIDA functional imaging scans.
Time Frame: 3 months
Population: The trial was halted prematurely because sponsor withdrew funding. There is insufficient data as funding to perform the analysis was withdrawn.
Arm/Group | MRI and HIDA Scan
Number analyzed (Participants) | 0

2. Secondary Outcome: Secondary
Description: Determine the difference in global liver function between pre and 3 months post Yttrium 90 delivery using the HIDA functional imaging scans.
Time Frame: 3 months
Population: The trial was halted prematurely because sponsor withdrew funding. There is insufficient funding for data to be analyzed properly.
Arm/Group | MRI and HIDA Scan
Number analyzed (Participants) | 0

3. Secondary Outcome: Secondary
Description: Correlation between the differences in liver function (both regional and global) with the Y 90 dose provided.
Time Frame: 6 months
Population: The trial was halted prematurely because sponsor withdrew funding. There is insufficient funding to properly analyze.
Arm/Group | MRI and HIDA Scan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | MRI and HIDA Scan
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
The trial was halted prematurely because sponsor withdrew funding. There is insufficient data to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT02966223/Prot_SAP_001.pdf